CLINICAL TRIAL: NCT02558764
Title: Effects of Preventive Negative Pressure Wound Therapy With PICO on Surgical Wounds of Kidney Transplant Patients: A Pilot Trial
Brief Title: Effects of Preventive Negative Pressure Wound Therapy With PICO on Surgical Wounds of Kidney Transplant Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Dr. Alwayn is leaving NSHA and Canada for a new appointment in Europe
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2015-09-18; First posted 2015-09-24 (Estimated); Last update posted 2022-10-28 (Actual); Status verified 2015-09

CONDITIONS: Wound Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): No intervention; basic wound contact absorbent dressings will be used as per current standard of care.
- PICO (Other): PICO device will be used for prevention of wound complications. This is a portable negative pressure wound treatment device. Patients will have the device for 7 days after undergoing kidney transplant surgery.
  Interventions: Device: portable (pocket) negative pressure wound treatment device

INTERVENTIONS:
Device: portable (pocket) negative pressure wound treatment device — PICO device will be applied to the surgical wounds of kidney transplant patients who are enrolled in the PICO group. These patients will have this device on for 7 days after undergoing kidney transplant surgery.
  Other Names: PICO, Smith & Nephew, London UK
  Arms: PICO

SUMMARY:
Advances in surgical techniques and immunosuppression (IS) have led to an appreciable reduction in postoperative complications following kidney transplantation. However, surgical site events (SSE) including surgical site infections (SSI) and other wound complications are still very common and they can limit these improved outcomes and result in prolonged hospitalization, hospital readmission and reoperation, consequently increasing overall transplant cost.

Negative pressure wound therapy (NPWT) is a concept introduced initially to assist in the treatment of chronic open wounds. This technique uses a negative pressure unit and specific dressings that help to hold the incision edges together, redistribute lateral tension, reduce edema, stimulate perfusion and protect the surgical site from external infectious sources. Thus, it provides faster wound healing and shortens hospital stay.

Recently, there has been growing interest in using portable NPWT devices on closed incisions after surgery to prevent potential SSI and other wound complications in high-risk patients. Investigations regarding this technique in various surgical settings have shown that it can reduce the risk of SSI and other wound complications. These studies concluded that any patient undergoing transplantation should be considered as 'high-risk' and should receive this treatment.

To date, no studies are reported in literature exploring the effects of preventive use of portable NPWT devices on surgical wounds in the setting of organ transplantation. The aim of our study is to compare a portable NPWT device (PICO, Smith & Nephew, London UK) to conventional gauze dressings in patients undergoing kidney transplantation (KT) surgery.

DETAILED DESCRIPTION:
Patients admitted to our transplant surgery inpatient floor for cadaveric kidney transplant surgery will be reviewed with the circle of care team and approached for consent if deemed suitable for this trial. A Nova Scotia Health Authority Research Ethics Board approved informed consent form will be utilized in the consent discussion and patients will be provided time to read the document in full before being asked for a decision on participation.

Patients who give their consent for the study will be randomized to 'PICO' or 'Control' group. The randomization process will be held during the time period between the admission of the patient to the inpatient floor and referral of the patient to the operating room. Randomization process will be conducted by the transplant fellow or the research associate who will randomly pick an envelope from a box full of 60 same-sized, same-colored and closed envelopes each time a patient gives consent. Among those 60 envelopes 30 will have the 'PICO' card inside, while the remaining 30 envelopes will have 'control' card. Assignment process will be completed when 30 consecutive patients are included in each group. There will be 1 control per case.

For both patient groups the surgical wound closure procedure will be the same: At the end of each cadaveric kidney transplant procedure the wound edges will be approximated by means of running subcuticular suture with non-absorbable stitches (3/0 polypropylene/polyethylene). For patients randomized to the 'PICO' group, PICO will be applied in the operating room immediately after closure and the continuous negative pressure set at -80 mmHg.

For patients randomized to the control group standard of care basic wound contact absorbent dressings will be applied in the operating room immediately after the closure of the surgical wound.

Follow-up care:

Control Group patients will have the surgical site dressing changed sterilely when too wet, and then removed after 48 hours post op. At this time the wound will be left exposed if no complications occur.

PICO group patients will keep the device in place for 7 days, and then have it removed on post-operative day 7. PICO Dressing replacement will be performed in cases where the dressing becomes too wet before day 7.

All patients will receive antibiotic prophylaxis 60 minutes before surgery as per our routine protocol: Cefazolin (1-2 gram) IV will be given as the first-choice antibiotic. Clindamycin (600-900 mg) IV will be given to penicillin-allergic patients.

Data regarding following parameters will be collected for each recipient: Age at the time of transplant surgery, gender, diabetic status, pre-transplant dialysis status (preemptive/hemodialysis/peritoneal dialysis), body mass index/ pre-transplant weight, pre-operative serum albumin level, Human Leukocyte Antigen (HLA) mismatch status, panel reactive antibody (PRA) , functional status of the graft (immediate graft function / delayed graft function) and in-hospital stay.

Following variables regarding KT surgery and allograft will be collected: Date of KT surgery, donor age, cadaveric donor type (brain death/cardiac death), cold ischemia time, warm ischemia time and operative time.

SSE will be evaluated on post-operative days 3, 7 and 30. Data on minor and major wound complications (superficial wound dehiscence, evisceration, seromas, incisional hernias, wound infections and wound necrosis) collected over the first 30 postoperative days will be recorded on follow-up forms by the same researcher. These data will include information regarding the type of the wound complication, whether or not an intervention was required and type and number of the interventions (therapeutic vacuum-assisted closure, percutaneous drainage and re-operation).

PICO and conventional dressing (control) groups will be compared in terms of afore-mentioned "wound complication risk factors" and descriptive "recipient, donor and allograft" parameters. Subsequently, investigators are planning to proceed with comparison of the outcomes among these two groups. Statistical analysis methods described below will be used for comparison of the groups in terms of the rates of wound complications and wound complication-related intervention and re-operation rates.

8. STATISTICAL ANALYSIS A) Power calculation There will be 1 control assigned per case. Prior data indicate that the failure (wound complication) rate among controls is 0.25. Findings of the previous studies regarding preventive PICO application correspond to a true relative risk of 2.5. Relevant power calculation analysis suggests assignment of 26 experimental and 26 control subjects ((to be able to reject the null hypothesis that relative risk equals 1 with probability (power) 0.8)).

The Type I error probability associated with this test of this null hypothesis is 0.05. An uncorrected chi-squared statistic will be used to evaluate this null hypothesis.

B) Analysis of data Results will be expressed as mean ± standard deviation. Categorical data will be compared using 2-tailed Fisher's exact test or Chi-squared test. Continuous variables will be compared using Mann-Whitney test. p < 0.05 will be considered statistically significant. Statistical analyses will be performed with computer software (SAS for Windows, version 9.2).

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years of age)
2. female/male cadaveric kidney transplant recipients who have a preoperative order for standard induction immunosuppression protocol (basiliximab and methylprednisolone) and give written consent will be included in this study.

Exclusion Criteria:

1. Patients who have a pre-operative order for a non-standard induction immunosuppression regimen
2. Patients deemed not capable to take care for the PICO device
3. Multi-organ transplant recipients (simultaneous liver-kidney transplant, simultaneous kidney-pancreas transplant)
4. Dual KT recipients (simultaneous kidney-kidney transplant)

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2017-03-10 (Actual); Study Completion 2017-03-10 (Actual)

PRIMARY OUTCOMES:
post-kidney transplant wound complication rates | up to 12 months
  Primary outcome of this study will be 'post- KT wound complication (superficial wound dehiscence, evisceration, seromas, incisional hernias, wound infections and wound necrosis) rates'. The potential relation of these complications with PICO application will be assessed.